CLINICAL TRIAL: NCT03277807
Title: Effect of Physical Activity in Pregnancy on Low Grade Inflammation: a Pilot Study
Brief Title: Physical Activity in Pregnancy
Acronym: PAP
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: EK 24-245 ex 11/12
Record Dates: First submitted 2017-08-31; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Pregnancy, Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — maternal venous blood (serum /plasma), cord blood (serum /plasma); placenta tissue (RNA later);
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active: pregnant women who are physically active (spend a minimum of 150min/week with moderate to vigorous physical activity)
- Inactive: pregnant women who are physically inactive (spend less than 150min/week with moderate to vigorous physical activity)
- risk for hypertensive disorders: pregnant women with a history of preeclampsia or positive history for metabolic conditions increasing the risk of hypertensive disorders in pregnancy

SUMMARY:
This prospective observational study assesses whether women who regularly exercise during pregnancy show reduced low grade Inflammation, compared to women who are not regularly exercising. Furthermore, the effects of regular physical activity in pregnancy on fetal and neonatal outcomes will be investigated. 3 groups of pregnant women will be formed (group 1: regularly physically active women; group 2: physically inactive women and group 3: women with a history of preeclampsia or positive history of metabolic conditions increasing the risk of hypertensive disorders in pregnancy).

DETAILED DESCRIPTION:
Pregnancy is a natural state of low grade inflammation in the mother and the feto-placental unit. The severity of this inflammation increases with higher pregravid Body Mass Index (BMI). This is reflected by an increase in pro-inflammatory cytokines in the maternal circulation and in the placenta. It has been proposed that the pro-inflammatory maternal and fetal environment plays a role in mediating pregnancy outcomes.

In non-pregnant individuals regular physical activity is associated with a reduced inflammatory state. The overall objective of the study is to investigate the interaction of maternal physical activity and pregnancy induced low-grade inflammation in the mother and feto-placental unit, and to assess th resulting effects on prenatal and postnatal development.

Specific research objective will be to study effects of maternal physical activity on:

1. low grade Inflammation in the mother an feto-placental unit;
2. maternal and fetal lipid profiles, including High Density Lipoprotein (HDL) proteome;
3. fetal growth and infant body composition;
4. transcriptomic and epigenetic profile in the placenta;
5. biomarkers of nutritive status;
6. psychological assessment: cardiac awareness; assessment of arterial stiffness; stress-coping questionaire

ELIGIBILITY:
Inclusion Criteria:

* ongoing pregnancy no later than 14 weeks of gestation
* giving informed consent

Exclusion Criteria:

* not wanting to give birth at the University Hospital
* gestational age > 14 weeks of gestation
* 3 or more consecutive miscarriages
* increased risk to or above 1:200 after combined test (Minimum parameters: maternal age, fetal crown-rump length (CRL), nuchal translucency, nasal bone and maternal biochemistry)
* fetal anomalies associated with possible growth or genetic anomalies
* Smoking
* diagnosed with Diabetes type 1 or 2 (T1D, T2D)
* for groups 1 and 2: maternal metabolic risk factors (autoimmune conditions, increased risk for thromboembolic events needing anticoagulative therapy)
* for groups 1 and 2: pre-pregnancy hypertension

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with an ongoing healthy pregnancy. 3 groups will be formed: Group1 consists of women performing moderate to vigorous physical activity (PA) before and in early pregnancy. Group2 consists of women who are not physically active, and Group3 consists of women with a risk of hypertensive disorders or metabolic diseases (not diabetes). PA before and in early pregnancy will be assessed with a screening questionnaire. Women reporting a minimum of 150 mins of moderate to vigorous PA per week will be classified as active, women with less PA will be classified as inactive. 20 women each group will be recruited not later than 14 weeks of gestation. Women will be recruited at the outpatient clinic at the Department of Obstetrics and Gynecology, Medical University of Graz.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2013-10-11 (Actual); Study Completion 2013-10-11 (Actual)

PRIMARY OUTCOMES:
low grade inflammation (in maternal and cord blood) | 1 year
  clinical inflammation markers: C-reactive protein, cytokines and chemokine (IL1b, IL1a, IL-2, IL-5, IL-6,IL-12, TNFa, MCP-1, MIP1-a) measured by ELISA and multiplexing arrays

SECONDARY OUTCOMES:
maternal and fetal (cord blood) lipid profiles | 1 year
  triglycerides, phospholipids, free fatty acids, HDL/LDL/total cholesterol
neonatal body composition (% body fat) | 1 year
  measured by air displacement plethysmography (Peapod)
maternal and newborn fat distribution | 1 year
  subcutaneous adipose tissue thickness at 15 defined body sites, measured by a lipometer
fetal growth | 1 year
  measured by ultrasound scanner
transcriptome of the placenta | 2 years
  measured by full genome arrays
epigenetic analysis of the placenta | 2 years
  analysed by 450k methylation arrays
biomarkers of nutritional status | 2 years
  measurement of blood levels of fatty acids (DHA, EPA, 15:0, 17:0), vitamin A, B1, B2, B6, D2/D3, C, E, homocysteine
psychological assessment | 1 year
  assessment of arterial stiffness, stress coping questionnaire, cardiac awareness

CONTACTS AND LOCATIONS:
Overall Officials: Bence Csapo, MD, Principal Investigator — Medical University of Graz